CLINICAL TRIAL: NCT05936931
Title: Developing a Young Adult-Mediated Intervention to Increase Colorectal Cancer Screening Among Rural Screening Age-Eligible Adults
Brief Title: Young Adult-Mediated Intervention to Increase Colorectal Cancer Screening
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left UF. Study transferring to VCU.
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HM20026698; R03CA270837-01A1 (NIH)
Record Dates: First submitted 2023-06-23; First posted 2023-07-10 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Young Adult-Mediated Intervention to Increase Colorectal Cancer Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aim 3: Single arm, open-label, pre-test/post-test design pilot trial (Other): Single arm, open-label, pre-test/post-test design pilot trial
  Interventions: Behavioral: Changes in CRC screening awareness and intentions

INTERVENTIONS:
Behavioral: Changes in CRC screening awareness and intentions — Using a single arm, open-label, pre-test post-test design (n=15 adult child/parent dyads), assess the impact of a young adult-mediated intervention to increase CRC screening among a paired age-eligible family member (e.g., parent/grandparent). The focus of the intervention will be on changes in CRC screening awareness and intentions among the age-eligible adult, but we hypothesize that the young adult could benefit as well. Thus, in addition to assessing feasibility and acceptability, we will assess changes in 1) CRC screening intentions among the age-eligible adults and 2) CRC health literacy and awareness of screening guidelines among the younger adult participant.

SUMMARY:
This study will garner preliminary data to develop a young adult-mediated intervention whereby a younger family member encourages their older family member to get colorectal cancer (CRC) screening. In Aim 1, survey data from n=150 younger (25-44 years old) and n=150 older (45-75 years old) adults living in rural communities will be collected. In Aim 2, intervention components will be evaluated using n=9 focus groups. The novel intervention will be assessed via a pilot trial (n=15 adult child/parent dyads) in Aim 3.

DETAILED DESCRIPTION:
Aim 1. Environmental Scan of Health Communications Landscape. Using quantitative methods, examine the health communications landscape of younger (25-44 years old) and older (45-75 years old) adults living in rural communities. N=300 survey responses (n=150 from each age group) will be analyzed to determine the primary channels and sources of health-related information, quantify the extent to which these residents engage in family communications about cancer screening, and identify potential strategies for upward communications. Individual factors (i.e., CRC screening knowledge, health literacy, and numeracy) and specific facilitators of and barriers to upward communication about CRC screening will be also assessed.

Aim 2. Message Development and Refinement. Using qualitative methods, develop and evaluate intervention components to facilitate effective upward communications about CRC prevention and screening. To accomplish this aim, we will: 1) use findings from Aim 1 to design intervention content and materials that leverage relevant communication channels and strategies, and address barriers to upward communication and 2) conduct n=9 focus groups with adult children 25-44 years of age (n=3), CRC screening age-eligible adults, 45-75 years old (n=3), and adult child/parent dyads (n=3), to assess message acceptability and refine key content areas. We will iterate and modify intervention components based on feedback.

Aim 3. Preliminary Testing. Using a single arm, open-label, pre-test post-test design (n=15 adult child/parent dyads), assess the impact of a young adult-mediated intervention to increase CRC screening among a paired age-eligible family member (e.g., parent/grandparent). The focus of the intervention will be on changes in CRC screening awareness and intentions among the age-eligible adult, but we hypothesize that the young adult could benefit as well. Thus, in addition to assessing feasibility and acceptability, we will assess changes in 1) CRC screening intentions among the age-eligible adults and 2) CRC health literacy and awareness of screening guidelines among the younger adult participant.

ELIGIBILITY:
Inclusion Criteria:

* Residents of counties in the Virginia/North Carolina CRC hotspot
* 25-75 years old
* Able to speak, write, and comprehend English
* Younger adult participants in Aims 3 must have an older, screening age-eligible relative with whom they speak with regularly (i.e., ≥ once every two weeks)

Exclusion Criteria:

• Participants in Aims 1 or 2 will be ineligible for Aim 3

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
CRC screening knowledge and awareness | 2-months post-intervention
  A composite index score on four awareness items and 14 knowledge items adopted from prior research
CRC screeningintentions | 2-months post-intervention
  A single item, based on previous CRC screening research

CONTACTS AND LOCATIONS:
Overall Officials: Carrie A Miller, PhD, MPH, Principal Investigator — Virginia Commonwealth University